CLINICAL TRIAL: NCT07148323
Title: HemoSphere Alta Clinical Development Study
Brief Title: HemoSphere Alta Study
Status: Recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-05
Record Dates: First submitted 2025-08-13; First posted 2025-08-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hemodynamic Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Primary Cohort (Swan): Up to 100 subjects with planned monitoring with a pulmonary artery catheter in the OR.
  Interventions: Device: HemoSphere Alta Monitor, Swan-Ganz IQ pulmonary arterial catheter, ForeSight IQ Large sensor, and Acumen IQ sensor

INTERVENTIONS:
Device: HemoSphere Alta Monitor, Swan-Ganz IQ pulmonary arterial catheter, ForeSight IQ Large sensor, and Acumen IQ sensor — Subjects with planned monitoring with a pulmonary artery catheter in the operating room, will be monitored with the above listed devices.

SUMMARY:
A prospective, non-randomized single arm study using the HemoSphere Alta Advanced Monitoring Platform and associated devices in adult subjects. Data collected from enrolled study subjects will be used for continual device development purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 18 years
3. Planned monitoring with a pulmonary artery catheter
4. Patient scheduled to undergo cardiac or liver transplant surgery lasting > 2 hours
5. Additional criteria for Sub-Cohort A (RVF)

   1. Possible Right Ventricular Dysfunction/Failure based on pre-operative assessment of previous Transthoracic Echocardiogram (TTE)
   2. Planned Transesophageal Echocardiogram (TEE) assessment during the operative procedure
6. Additional criteria for Sub-Cohort B (CAI)

   1. Age ≥ 45 years
   2. Planned cardiac surgery with Cardiopulmonary Bypass (CPB)
   3. Ability to place ForeSight IQ and Acumen IQ sensors during the operative monitoring period
   4. High risk for cerebral vascular disease, defined as: a history of hypertension, pulse pressure > 60 mmHg, diabetes, stroke, transient ischemic attack, carotid bruit, tobacco smoking, or peripheral vascular disease

Exclusion Criteria:

1. Inability to provide informed consent
2. Pregnancy as confirmed per EMR
3. Patients deemed not suitable for the study at the discretion of the Investigator
4. Participation in another study that clinically interferes with the current study
5. Additional exclusion criteria for Sub-Cohort A

   1. Presence of left bundle branch block
   2. Presence of current/recurrent sepsis
   3. Presence of hypercoagulability, as identified in the patient's past medical history and preoperative evaluation
   4. Structural abnormality, including congenital heart defects, of the right ventricle
6. Additional exclusion criteria for Sub-Cohort B a. Surgery for congenital heart defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 subjects with planned monitoring with a pulmonary artery catheter in the Operating Room (OR). Subjects must meet the eligibility criteria for the Primary Cohort to be enrolled in the study. Subjects may further qualify for inclusion in Sub-Cohorts A and/or B.
  Sub-Cohort A Right Ventricular Failure (RVF) will include up to 25 subjects undergoing either non-cardiac or cardiac surgery with a planned transesophageal echocardiogram (TEE) assessment.
  Sub-Cohort B Cerebral Autoregulation Index (CAI) will include up to 50 subjects aged ≥ 45 years undergoing Cardiopulmonary Bypass (CPB) with the ability to place ForeSight and Acumen IQ sensors and are at high risk for cerebrovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Data Collection using HemoSphere Alta Advanced Monitoring Platform and associated devices | Up to 72 hours of device data collection during surgery and ICU
  Number of patients who receive monitoring using the HemoSphere Alta Advanced Monitoring Platform and associated devices for continued device development.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No